CLINICAL TRIAL: NCT03842111
Title: American Indian and Alaska Native Head Start Family and Child Experiences Survey (AI/AN FACES)
Brief Title: American Indian and Alaska Native Head Start Family and Child Experiences Survey
Acronym: AI/AN FACES
Status: Completed | Type: Observational
Sponsor: Mathematica Policy Research, Inc. (Other)
Collaborators: Children's Bureau - Administration for Children and Families (Other); Tribal Early Childhood Research Center (Unknown); Department of Health and Human Services (U.S. Federal Agency); Office of Planning, Research & Evaluation (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 40290B
Record Dates: First submitted 2017-10-12; First posted 2019-02-15 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-02

CONDITIONS: Head Start Participation
Keywords: Alaska natives; child care; child development; child health; child rearing; children; curriculum; early childhood education; families; Head Start; Native Americans; parenting skills; parents; programs; school readiness; teachers

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Region XI Head Start children and families: children (1049) parents (1049) classrooms/teachers (73) program directors (21) center directors (36)

SUMMARY:
The Head Start Family and Child Experiences Survey (FACES) is a major source of information on Head Start programs and the children and families they serve. Since 1997, FACES has conducted studies in a nationally representative sample of Head Start programs, but has historically not included Region XI (programs operated by federally-recognized tribes), whose programs are designed to serve predominantly American Indian and Alaska Native (AI/AN) children and families. The American Indian and Alaska Native Head Start Family and Child Experiences Survey (AI/AN FACES), the first national study of Region XI AI/AN Head Start children and families, is designed to fill this information gap.

For more information on FACES, please refer to the ClinicalTrials.gov ID NCT03705377.

DETAILED DESCRIPTION:
The Head Start Family and Child Experiences Survey (FACES) is a major source of information on Head Start programs and the children and families they serve. Since 1997, FACES has conducted studies in a nationally representative sample of Head Start programs, but has historically not included Region XI (programs operated by federally-recognized tribes), whose programs are designed to serve predominantly American Indian and Alaska Native (AI/AN) children and families. The American Indian and Alaska Native Head Start Family and Child Experiences Survey (AI/AN FACES), the first national study of Region XI AI/AN Head Start children and families, is designed to fill this information gap.

The design of AI/AN FACES has been informed by members of the AI/AN FACES Workgroup which includes tribal Head Start directors, researchers with expertise working with tribal communities, Mathematica Policy Research study staff, and federal officials from the Office of Head Start, Region XI, and the Office of Planning, Research and Evaluation. Building on FACES as the foundation, members of the AI/AN FACES Workgroup have shared insights and information on the kinds of information needed about children and families served by Region XI AI/AN Head Start programs (including children's development and school readiness, parent and family demographics, health, and program engagement, and teacher, classroom, and program characteristics). Members also provided input on recruitment practices and study methods that are responsive to the unique cultural and self-governing contexts of tribal Head Start programs.

Data collection with Region XI children, families, classrooms, and programs took place in the Fall of 2015 and the Spring of 2016. Twenty-one Region XI Head Start programs participated. Procedures for tribal review and approval in each of those 21 communities were followed. Information about this study has been shared broadly with tribal Head Start programs and tribal leaders via Office of Head Start (OHS) tribal consultations, nationally-broadcast webinars, National Indian Head Start Directors' Association Board of Directors (NIHSDA) annual conferences, the 2016 Administration for Children and Families (ACF) National Research Conference on Early Childhood, and the Secretary's Tribal Advisory Council (STAC) December 2014 and 2016 meetings.

ELIGIBILITY:
Inclusion Criteria:

- The Region XI AI/AN Head Start programs participating in AI/AN FACES were a probability sample selected from among 147 study-eligible programs on the 2012-2013 Head Start Program Information Report (PIR). To be eligible for the study, a program had to be providing services directly to children ages 3 to 5, and not be in imminent danger of losing its grantee status. Probability samples of centers were selected within each program, classrooms within each center, and children within each classroom. Teachers associated with selected classrooms were included in the study with certainty, as were parents associated with selected children.

Exclusion Criteria:

- Head Start programs in Regions I through X and Migrant and Seasonal Head Start (Region XII) were not eligible for AI/AN FACES. Other ACF studies (FACES-NCT03705377 and MSHS-NCT03116243) focus on those programs.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Region XI Head Start children (and their families), Region XI Head Start programs, Region XI Head Start centers, Region XI Head Start classrooms/teachers
Sampling Method: Probability Sample
Enrollment: 1194 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
English proficiency | 1 year
  Children's English language proficiency was assessed during week-long site visits using Preschool Language Assessment Survey (preLAS 2000): Simon Says and Art Show. See Duncan and DeAvila for more information on the scores and technical properties.
  Duncan, S.E., and E. DeAvila. Preschool Language Assessment Survey 2000 Examiner's Manual: English Forms C and D. Monterey, CA: CTB/McGraw-Hill, 1998.
Language-English receptive vocabulary | 1 year
  Indicators of language were assessed during week-long site visits using Peabody Picture Vocabulary Test-Fourth Edition (PPVT-4). See Dunn and Dunn 2006 for more information on the scores and technical properties.
  Dunn, L. M., & Dunn, D. M. Peabody Picture and Vocabulary Test, Fourth Edition. Examiner's Manual and Norms Booklet. Circle Pines, MN: American Guidance Service, 2006.
Language-Expressive vocabulary | 1 year
  Indicators of language were assessed during week-long site visits using Expressive One-Word Picture Vocabulary Test-Fourth Edition (EOWPVT-4). See Martin and Brownell 2011 for more information on the scores and technical properties.
  EOWPVT-4: Martin, N., and R. Brownell. "Expressive One-Word Picture Vocabulary Test-4th Edition." Novato, CA: Academic Therapy Publications, 2011.
Literacy-Letter word knowledge/early writing | 1 year
  Indicators of literacy were assessed during week-long site visits using Woodcock-Johnson III Tests of Achievement-Third Edition (Spelling, Letter-Word Identification). Please see Woodcock et al. 2001 for more information on the scores and technical properties.
  Woodcock, R. W., McGrew, K. S. & Mather, N. (2001). Woodcock-Johnson III Tests of Achievement, Itasca, IL: Riverside Publishing, 2001.
Literacy-Letter sounds knowledge | 1 year
  Indicators of literacy were assessed during week-long site visits using ECLS-B Letter Sounds. Please see Snow et al. 2007 for more information on the scores and technical properties.
  Snow, K., L. Thalji, A. Derecho, S. Wheeless, J. Lennon, S. Kinsey, J. Rogers, M. Raspa, and J. Park. "Early Childhood Longitudinal Study, Birth Cohort (ECLS-B), Preschool Year Data File User's Manual (2005-06)." NCES 2008-024. Washington, DC: National Center for Education Statistics, Institute of Education Sciences, U.S. Department of Education, 2007.
Mathematics | 1 year
  Indicators of mathematics were assessed during week-long site visits using the Early Childhood Longitudinal Study-Birth Cohort (ECLS-B) preschool mathematics assessment of children's understanding of relative size, ordinal numbers, and pattern matching; number recognition; and the children's ability to count, recognize shapes, add, and solve word problems. Please see Snow et al. 2007 for more information on the scores and technical properties.
  Snow, K., L. Thalji, A. Derecho, S. Wheeless, J. Lennon, S. Kinsey, J. Rogers, M. Raspa, and J. Park. "Early Childhood Longitudinal Study, Birth Cohort (ECLS-B), Preschool Year Data File User's Manual (2005-06)." NCES 2008-024. Washington, DC: National Center for Education Statistics, Institute of Education Sciences, U.S. Department of Education, 2007.
Mathematics | 1 year
  Indicators of mathematics were assessed during week-long site visits using the Woodcock-Johnson III Tests of Achievement-Third Edition (Applied Problems Test). Please see Woodcock et al. 2001 for more information on the scores and technical properties.
  Woodcock, R. W., McGrew, K. S. & Mather, N. (2001). Woodcock-Johnson III Tests of Achievement, Itasca, IL: Riverside Publishing, 2001.
Children's physical health | 1 year
  Indicators of physical well-being were assessed by weighing (using kilograms) and measuring children's height (using centimeters), and using these measurements to calculate Body Mass Index (BMI).
General health status | 1 year
  Indicators of physical well-being were assessed by parent report to a survey item on if child's health is excellent, very good, good, fair, or poor.
Executive function | 1 year
  Indicators of executive function were assessed by a pencil-tapping task that requires the child do the opposite of what the assessor says (that is, tap one time when the assessor taps two times and tap two times when the assessor taps one time). Pencil Tapping provides an objective assessment of children's self-regulation, particularly inhibitory control and working memory.
  See Blair 2002 for example for more information on the task.
  Blair, C. "School Readiness: Integrating Cognition and Emotion in a Neurobiological Conceptualization of Children's Functioning at School Entry." American Psychologist, vol. 57, 2002, pp. 111-127.
Social-emotional development | 1 year
  Indicators of social-emotional development were assessed using teacher report of several items on children's positive and problem behaviors. Please see the AI/AN FACES 2015 User's Manual (Malone et al. 2018) for more information on the scores and technical information.
  Malone, L., A. Kopack Klein, S. Bernstein, B. Carlson, S. Albanese, A. Bloomenthal, J. Baker, M. Cavanaugh, M. Reid, K. Feeney, R. Sutton-Heisey, M. Hepburn, A. Kelly, and G. Lim. "American Indian and Alaska Native Head Start Family and Child Experiences Survey 2015 (AI/AN FACES 2015) User's Manual." Report submitted to the U.S. Department of Health and Human Services, Administration for Children and Families, Office of Planning, Research, and Evaluation. Washington, DC: Mathematica Policy Research, 2018.
Social-emotional development-cognitive/social behaviors | 1 year
  Indicators of social-emotional development were assessed using assessor report children's cognitive/social behaviors during the assessment time, using the Leiter-R Examiner Ratings. The Leiter-R comprises eight subscales that examine children's approach to the assessments, their engagement with the materials, and their ability to attend to and regulate their physical and emotional responses during the assessment tasks. Please see Roid and Miller 1997 for more information on the scores and technical properties.
  Roid, G.H., and L.J. Miller. Leiter International Performance Scale Revised, Examiner Rating Scale (Leiter-R). Lutz, FL: Psychological Assessment Resources, Inc., 1997.
Social-emotional development - Approaches to learning | 1 year
  Indicators of social-emotional development were assessed using teacher report of approaches to learning using the Early Childhood Longitudinal Study - Kindergarten Class of 1998 (ECLS-K). The items assess a child's motivation, attention, organization, persistence, and independence in learning. Please see U.S. Department of Education 2002 for more information on the scores and technical properties.
  U.S. Department of Education, National Center for Education Statistics. "Early Childhood Longitudinal Study-Kindergarten Class of 1998-99 (ECLS-K), Psychometric Report for Kindergarten through First Grade." NCES 2002-05. Washington, DC: National Center for Education Statistics, Institute of Education Sciences, U.S. Department of Education, 2002.
Classroom quality-teacher child interactions | One-day observation in March-May 2016
  Indicators of classroom quality were assessed using the the PreK Classroom Assessment Scoring System. The Pre-K CLASS assesses the qualities of interactions between teachers and students in classrooms and measures aspects of interactions related to children's early academic achievement and social competencies. Please see Pianta et al. 2008 for more information on the scores and technical properties.
  Pianta, Robert, K. LaParo, and B. Hamre. The Classroom Assessment Scoring System Pre-K Manual. Charlottesville, VA: University of Virginia, 2008.
Classroom quality-global classroom environment | One-day observation in March-May 2016
  Indicators of classroom quality were assessed using a shortened form of the Early Childhood Environment Rating Scale-Revised (ECERS-R), a global rating of classroom quality based on structural features of the classroom (Harms et al. 2005). The items in the short form represent the strongest 21 items identified by researchers in a large-scale study (Clifford et al. 2005). Please see Harms et al. 2005 and Clifford et al. 2005 for more information on the scores and measure technical properties.
  Harms, T., R.M. Clifford, and D. Cryer. Early Childhood Environment Rating Scale: Revised Edition. New York: Teachers College Press, 2005.
  Clifford, Richard, Oscar Barbarin, Florence Chang, Diane M. Early, Donna Bryant, Carollee Howes, Margaret Burchinal, and Robert Pianta. "What Is Pre-Kindergarten? Characteristics of Public Pre-Kindergarten Programs." Applied Developmental Science, vol. 9, no. 3, 2005, pp. 126-143.
Classroom quality-Native cultural and language experiences | One-day observation in March-May 2016
  Indicators of Native culture and language were assessed using Included a cultural items checklist on the presence and use of items such as cultural and Native language books or Native musical instruments, and a set questions on whether storytelling occurred, whether a tribal language was used, and whether any other activities exposed children to tribal culture during the observation.

CONTACTS AND LOCATIONS:
Overall Officials: Lizabeth Malone, Ph.D., Study Director — Mathematica Policy Research; Nikki Aikens, Ph.D., Principal Investigator — Mathematica Policy Research; Louisa Tarullo, Ed.D., Principal Investigator — Mathematica Policy Research
Locations (1):
- Mathematica Policy Research, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Yes
The AI/AN FACES study team prepared a restricted-use data file and documentation so that future researchers may use the data to replicate findings and explore new areas of inquiry.
Supporting Information: Study Protocol
Time Frame: Data are available for AI/AN FACES 2015 at ResearchConnections.org.
Access Criteria: Access to AI/AN FACES 2015 data is limited to individuals working in institutions of higher education or research organizations. In addition to completing the Inter-university Consortium for Political and Social Research (ICPSR) standard application, researchers must complete additional requirements in order to obtain access to the AI/AN FACES 2015 data.
URL: https://www.researchconnections.org/childcare/studies/36804

REFERENCES:
- See also: To learn more about AI/AN FACES and access reports/publications, please visit the AI/AN FACES ACF website. — https://www.acf.hhs.gov/opre/research/project/american-indian-and-alaska-native-head-start-family-and-child-experiences-survey-faces
- See also: To learn more about AI/AN FACES and access reports/products, you may also visit the Mathematica study website. — https://www.mathematica-mpr.com/our-publications-and-findings/projects/american-indian-and-alaska-native-head-start-family-and-child-experiences-survey-ai-an-faces